CLINICAL TRIAL: NCT03545048
Title: A Randomized Controlled Trial Evaluating the Efficacy of Internet-Based Exercise Program Aimed at Treating Knee Osteoarthritis (iBEAT-OA)
Brief Title: Effects of Internet / Web-based Exercises on the Population With Knee Arthritis
Acronym: Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Arthritis Research UK (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Sameer Gohir, PhD student, Extended Scope Practitioner, MSK sonographer, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 18021
Record Dates: First submitted 2018-05-01; First posted 2018-06-04 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Sleep Disturbance
Keywords: web-based exercises; Digital health; knee exercises
MeSH Terms: conditions — Osteoarthritis, Knee; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Interventional groups will have an assessment session with the experienced staff and NRS, QST, WOMAC, MSK-HQ, 30CST, TUG, PSQI, MSK-USS, urine and blood samples will be taken at baseline. Those who consent for aspiration of synovial fluid will go through the USGA procedure.
  Interventional group will shortly after that receive a link via email, which will be used to log-in to Joint Academy online portal. After log-in has been achieved, the intervention starts. It consist of a 6-week internet-based physical therapy program. Interventional group will be given actigraphy device (a device to monitor sleeping pattern) which is CE marked. Therefore, their sleeping pattern can be recorded quantitatively.
  Once exercises programme is finished in six weeks, the participants will fill in the same questionnaire and perform the physical tests, to enable evaluation.
  Interventions: Other: Internet based exercises
- Control arm (No Intervention): Control group will continue with their routine self-management which is offered in the community setup. They will be assessed on NRS, QST, WOMAC, MSK-HQ, PSQI, 30CST, TUG, isometric muscles strengthen of quadriceps, MSK-USS, muscle mass of vastus lateralis, urine and blood samples at baseline. Control group will also get the actigraphy to monitor sleeping pattern of that group. They will be re-assessed after six weeks on the primary objective measures to see if they have made any difference by following self-management strategies in the community.

INTERVENTIONS:
Other: Internet based exercises — Exercises for knee OA (online- digital health)
  Arms: Intervention arm

SUMMARY:
1. To test whether internet-based exercises reduce the pain in knee OA
2. To check whether internet-based exercises improve the physical activity in the patients with knee OA.
3. To explore the correlation between sleep, knee inflammation (effusion, synovial hypertrophy or/and synovial hyper vascularity) and biomarkers of insulin resistance and knee pain.

DETAILED DESCRIPTION:
Osteoarthritis is the most common cause of disability in the elderly population and most individuals suffering from osteoarthritis is managed in the primary care setting (1). Knee osteoarthritis is a most common form of arthritis in the world (2). The rate of knee arthritis is as high as that of cardiac disease and is the most common problem in the individuals over the age of 65 (3). In the United Kingdom, 10% of 65-74-year-old individuals consult their general practitioners about osteoarthritis per year (4). 4% population attend their general practitioners as a result of knee osteoarthritis and half of them (2%) consult their general practitioner for the first time or with the acute flare of knee arthritis (1).

According to national and international guidelines, the first line treatment for osteoarthritis pain (OA) is non-surgical; exercise, information and, in relevant cases, weight loss (5-9). There is enough evidence for the effectiveness of exercises in the management of knee osteoarthritis and to improve the functional capacity of these individuals to cope better with the activities of daily living (10-24). In fact, one study reported a slow down of progressive radiographic changes of knee OA as a result of strengthening exercises (25).There is a significant disparity on the effectiveness of different types of exercises for the knee osteoarthritis, and a combination of open and closed isotonic exercises are recommended knee osteoarthritis (26) with the exception to those individuals who find these exercises difficult and painful. In such groups, isometric exercises of knee muscles should be considered (26). In an attempt to manage the knee osteoarthritis, one can exacerbate the symptoms of knee arthritis by following ineffective or unsafe exercises leading to poor prognosis and poor adherence to these exercises (27), hence one should choose the exercises carefully.

As knee arthritis is a significant issue in the elderly population, therefore, the less expensive community-based approach will be beneficial for these patients. There are previous studies which have assessed the efficacy of home-based exercises and reported good results (12, 14, 28) however there are only a few studies which looked at the web-based exercises on the knee arthritis (29-33). Unfortunately, most of these studies recruited patients with knee pain, and radiographic evidence of knee osteoarthritis was undermined except one study (31). It infers that these web-based exercises can be used for knee pain which may include cases of soft tissue injuries, arthritic knee or any other reason for knee pain. However, generalising these results on the group of patients with knee osteoarthritis warrants a risk of increasing their pain just in case that those exercises are strenuous or more demanding.

The aim of this study is to explore the benefits of web-based exercises in the patients with knee osteoarthritis to establish if their pain decreases after six weeks. Being a web-based set of activities, it makes it more accessible to the patients living in rural areas and should make it more cost-effective requiring no travelling time. Our study is different from the other studies as there is not a single study (to our knowledge) which has studied web-based intervention on United Kingdom population of knee osteoarthritis. Furthermore, the investigators will endeavour to recruit only those individuals who have radiographic evidence of knee osteoarthritis. Therefore, this study will produce recommendations for the clinical setups where most of the symptomatic patients have radiographic evidence of knee osteoarthritis. The investigators will be using a web-based exercises platform known as Joint Academy (JA) as recent pilot studies (32, 33) demonstrated promising results for this platform. This programme is based on Swedish face to face self-management program known as 'Artrosskolan' (The Osteoarthritis School) which provides structured information and exercises for knee arthritis to the relevant population suffering from knee arthritis. The efficacy of it is covered elsewhere (34). The company that produced the Joint Academy platform has given consent to use their web based platform to conduct this study.

The investigators will recruit 134 individuals with the clinical evidence of radiographic knee arthritis, and these will be randomised into a control group and an interventional group (67 individuals in each group). The interventional group will get the login details for the Joint Academy (JA), and they will follow the strengthening exercises for six weeks with educational material online relevant to knee osteoarthritis. They will record their pain levels on the Numerical rating scale (NRS) at baseline and at the end of the trial. The validity and sensitivity of NRS have been established numerous times (35-39). Other than determining the subjective pain levels, the investigators will use standardised quantitative sensory testing (QST) such as pressure pain threshold (PPT), temporal summation (TS) and conditioned pain modulation (CPM). Pressure Pain threshold (PPT) has been used in previous studies done on the knee arthritis and deemed to be a valid and reliable method to establish tenderness around the knee joint (40-45). Similarly, temporal summation (TS) has been used in previous studies (40, 43, 44, 46) to establish whether individuals have an element of central sensitisation thus amplifying their localised knee pains. Conditioned pain paradigms are commonly used to assess the function of endogenous pain inhibitory pathways in humans. In this technique, a painful test stimulus is evaluated in the absence and in the presence of a second painful (conditioning) stimulus applied to a remote region of the body. In a typically functioning nociceptive system, the amount of pain experienced with the primary test stimulus will be reduced during the presentation of the secondary conditioning stimulus (47-49). Decreased inhibition of experimental pain is found in many patients with idiopathic pain syndromes (50-58). It predicts the tendency to develop future chronic pain (59, 60). The purpose of using QST is to establish objective data as to whether these exercises reduce the localised tenderness or global central sensitisation.

The investigators will use the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) which is widely utilised in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire made of 24 items and consists of three subscales covering pain, stiffness and physical function. It has been used extensively and deemed to be a valid and reliable tool (61-65). For the quality of life, stiffness, generalised well-being, difficulty with sleeping and understanding of the diagnosis and treatment, the investigators will use patient-reported outcome measure 'The Arthritis Research UK Musculoskeletal Health Questionnaire' (MSK-HQ). MSK-HQ covers a broad aspect of musculoskeletal conditions, and recent studies have shown it to be reliable and valid (66, 67).

Both the 30-second sit to stand test (30CST) and the 'time up and go' (TUG) test will be used to see if you have improved their lower limb fitness levels. 30CST has shown excellent reliability and validity (65, 68, 69). TUG has been widely used in clinical setups and is a valid tool to assess necessary functional mobility (70-76).

In this study, the investigators aim to assess the sleeping pattern of individuals suffering from degenerative changes of the knee and purpose is to determine whether sleeping patterns improve when the exercises for knee osteoarthritis are introduced. Disturbed sleep is a frequent complaint of people experiencing chronic pain such as those with knee osteoarthritis (OA) (77-83). The resultant changes in sleep architecture can affect health even in the presence of apparently adequate sleep duration. For example, an insufficient amount of slow wave sleep associates with hypertension, type 2 diabetes mellitus, poor cognition and obesity (84-89).Sleep disturbances are present in 67-88% of people with chronic pain and ≥50% individuals with insomnia have chronic pain (85, 90). Actigraphy will be used to assess the sleeping data which has been used widely and deemed as a valid method (91-96). The investigators will also use Pittsburgh sleep quality index (PSQI) which has been used in multiple studies and validated to measure sleep disturbances (97-101).

The investigators aim to conduct Musculoskeletal Ultrasound scan (MSK-USS) on the knees of these individuals to establish if they have inflammation of synovial membrane. There is enough evidence that inflammation is present in all stages of osteoarthritis (102-105). Synovitis or inflammation of synovial fluid is associated with pain, disease severity and progression of osteoarthritis (102, 106). Synovitis manifests as synovial membrane thickening, increased vascularity and/or joint effusion (102, 107-109). As standard radiographs are unable to visualise the synovial membrane, therefore, the investigators anticipate using an ultrasound machine. The investigators will assess synovial fluid, hypertrophy of synovium and presence of Power Doppler during the ultrasound scan. Synovial hypertrophy, synovitis and knee effusion are linked with arthritis in the knee and associated with knee pain in osteoarthritis (110-115). Power Doppler provides a reliable and accurate method for visualising blood flow in the synovial tissue, and histological findings support the value of this technique (113, 116, 117). An ultrasound scan is proved to be a valid and reliable instrument for the assessment of synovial disease (107, 113, 114, 118) and synovitis is strongly associated with osteoarthritis as mentioned earlier. The investigators aim to aspirate the synovial fluid (SF) (subjective to the consent of the patient), and the purpose is to establish if the investigators can assess the synovial fluid to predict the phenotype which is strongly associated with osteoarthritis. Studying synovial fluid (SF) biomarkers alongside clinical, radiographic and ultra-sonographic characteristics is one strategy to improve resolution and stratification into targetable OA phenotypes (119). Ultrasound-guided aspiration (USGA) of synovial fluid is a safe procedure and less painful when compared to anatomical guided aspirations (120-123).

The investigators will also endeavour to assess the isometric strength of quadriceps to establish if these exercises improve the dynamic strength of knee extensors. Quadriceps muscles strength deficits are associated with knee osteoarthritis (124). Isometric testing will be done at 30 and 60 degrees of flexion as done in a previous study (125).

The investigators aim to ultrasound the muscle mass around the knee and wishes to check if six weeks exercise program results in any difference to the muscle mass around the knee. There are conflicting results whether vastus medialis or vastus lateralis atrophies significantly when all four muscles of quadriceps have been assessed and compared. It is evident that decreased strength of quadriceps muscles is found in the population suffering from the knee arthritis (126-130). One study suggested that all four muscles of knee extensors atrophy similarly in the elderly population (131). Another study reported atrophy of type 2 fibres in vastus lateralis and associated it to osteoarthritis when compared to controlled group (132). Other studies have associated atrophy of vastus medialis with arthritis (133, 134) and greater vastus medialis cross-sectional area is associated with reduced knee pain and reduced medial tibial cartilage loss (135). A recent study has studied the sonographic changes of vastus lateralis after introducing exercises and correlated the findings to the MRI scan, and they conclude that ultrasound is a valid method of assessing muscle thickness (136). This study has used vastus lateralis muscle to conclude these findings and therefore the investigators plan to measure vastus lateralis muscle mass thickness and pennation angle as described in earlier studies (136, 137). The pennation angle is defined as the angle between muscle fibres and the deep fascia of the muscle (137). The pennation angle correlates with the maximum voluntary contraction (MVC) force which is a measurement of muscle strength (137), thus the ultrasound scan will indirectly establish if the exercises have led to an increase in maximum voluntary contraction.

The investigators will also extract the blood samples at baseline and after six weeks to assess the biomarkers and to establish insulin resistance (138, 139). A urine sample will be taken as well.

Studying these parameters will help us to understand the traits of osteoarthritis, their correlation to each other and potential detrimental effects of them on the health of knee joint. This study will help us to establish whether web-based intervention can replicate the results which it has produced in Swedish population and if it does, then next target will be to assess the socio-economic benefits of this programme over the standard treatment for knee arthritis provided in the community set up in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 years and onward.
* Clinical diagnosis of knee arthritis with complaints of knee pain for 3-6 months, early morning stiffness <30 minutes, crepitus, bony tenderness, and no palpable warmth and radiographically established osteoarthritis (at least score 1 on K/L scale)
* Able to read and write English
* Able to use/access computer or tablet and have access to internet

Exclusion Criteria:

* Inability to give informed consent - (capacity levels are already established under General practitioner care)
* Terminal or mental illness
* Neurological conditions, inflammatory joint diseases including rheumatoid arthritis, gout or calcium pyrophosphate deposition disease (CPPD), and dementia
* Patients with sleep apnea
* Acute soft tissue injury to the knee within last 3 months before recruiting
* Unstable heart condition or rapid fluctuations in hypertension

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Knee pain measured on Visual Analogue Scale | 6 weeks
  knee pain scored on 00- 10 (00 no pain and 10 being worst pain)

SECONDARY OUTCOMES:
Pittsburgh sleep quality index (Sleep disturbances ) | 6 weeks
  Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Quantitative Sensory Testing (Pressure pain threshold - PPT) | 6 weeks
  PPT is a non-invasive test during which the sensitivities of the nerves are assessed by recording the smallest force applied to the skin. When this force by the surface area of the skin is applied (pressure), this will be felt as mild, temporary pain and recorded. The pressure probe used consists of a rod with an end the size of a 5p piece, mounted in a handheld device connected to a computer. The force with which the probe is pressed onto the skin is gradually increased until the participant indicates (by pressing a button) that the sensation has changed from pressure to pain. The probe is then automatically immediately taken off the skin.
Ultrasound of the knee | 6 weeks
  During the ultrasound scan, the maximal synovial thickness and effusion depth will be measured in millimetres using the longitudinal axis. Suprapatellar pouch, medial and lateral recess of the knees will be assessed for synovial thickening, synovial fluid/effusion and for positive power Doppler.
Muscle mass on musculoskeletal ultrasound | 6 weeks
  Muscle mass of Vastus Lateralis
The Timed Up and Go test (TUG) | 6 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
  One source suggests that scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Western Ontario and McMaster Universities Osteoarthritis Index | 6 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
General health questionnaire (MSK-HQ) | 6 weeks
  MSK-HQ is indicative of an overall rating of a person's musculoskeletal health at any given time; the MSK-HQ enables patients and their clinicians to monitor progress over time and response to treatment.
  Followings are assessed on MSK-HQ;
  * pain severity (in the day and night),
  * physical function (walking and dressing),
  * physical activity level,
  * pain interference (with work/daily routine and with social activities/hobbies),
  * difficulty with sleep, fatigue/low energy levels,
  * emotional well-being (anxiety and mood),
  * understanding of diagnosis and treatment,
  * confidence to self-manage (pain self-efficacy),
  * independence,
  * overall impact from symptoms (bothersomeness).
  There are 14 questions on MSK-HQ and participants are check pre and post intervention to see if they have made any difference due to intervention.
The 30 seconds sit to stand test | 6 weeks
  The 30CST is a measurement that assesses functional lower extremity strength in older adults. The 30-second chair stand involves recording the number of stands a person can complete in 30 seconds rather than the amount of time it takes to complete a pre-determined number of repetitions. A healthy male of 60-64 year old should be able to complete 17 sit to stand in 30 seconds whereas female of similar age should be able to complete 15 sit to stand.
Continuous Pain Modulation (CPM) | 6 weeks
  CPM will be done along with PPT testing. In this test, an external painful stimulus is introduced to check whether new stimulus reduces or amplifies the pain which is being studied. A blood pressure cuff is used and pain target will be 4 out of 10 from the cuff pressure.
  Once NRS of 4 will be achieved, the probe of algometer will be applied in the same manner as before to knee test site (during PPT testing). Once the participant presses the button, the probe will be withdrawn, and cuff will be released from the elbow.
  Participants will be advised to wait until cuff evoked pain subsides before re-test, and a minimum of 1 minute should be spared. PPT test will be repeated again (without the cuff now). Their difference in PPT score (with conditioning - without conditioning) will establish the CPM effects. Positive value predicts efficient and negative value predicts in-effective CPM.
Temporal Summation (TS) | 6 Weeks
  The mechanical temporal summation is a non-invasive test during which repetitive mechanical stimulation is applied over a short period to get their augmented response. Increased pain response to a repeated mechanical stimulus may indicate enhanced central sensitisation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, East Midland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gohir SA, Eek F, Kelly A, Abhishek A, Valdes AM. Effectiveness of Internet-Based Exercises Aimed at Treating Knee Osteoarthritis: The iBEAT-OA Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e210012. doi: 10.1001/jamanetworkopen.2021.0012. PMID 33620447
- [Derived] Gohir SA, Greenhaff P, Abhishek A, Valdes AM. Evaluating the efficacy of Internet-Based Exercise programme Aimed at Treating knee Osteoarthritis (iBEAT-OA) in the community: a study protocol for a randomised controlled trial. BMJ Open. 2019 Oct 28;9(10):e030564. doi: 10.1136/bmjopen-2019-030564. PMID 31662373